CLINICAL TRIAL: NCT01015638
Title: Two-week Study to Determine and Compare the Tolerance and Irritation Potential of Duac® Topical Gel (Clindamycin 1% and Benzoyl Peroxide 5%) to ACANYA™ Gel (Clindamycin Phosphate 1.2% and Benzoyl Peroxide 2.5%) Topical Acne Medications
Brief Title: Compare the Tolerance of Clindamycin 1% /Benzoyl Peroxide (BPO) 5% Gel to Clindamycin 1.2%/ BPO 2.5% Topical Medications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 114546
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2012-02-13 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Acne Vulgaris
Keywords: Healthy volunteers
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin; Gels; clindamycin phosphate; Benzoyl Peroxide; Acanya Gel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clindamycin and BPO 5% gel (Experimental): Once-daily applications, to the randomized side of the face either left or right, of clindamycin and benzoyl peroxide (BPO) 5% gel.
  Interventions: Drug: Clindamycin and BPO 5% gel
- Clindamycin phosphate and BPO 2.5% gel (Active Comparator): Once Daily application of clindamycin phosphate and benzoyl peroxide (BPO) 2.5% gel.
  Interventions: Drug: Clindamycin phosphate and benzoyl peroxide 2.5% gel.

INTERVENTIONS:
Drug: Clindamycin and BPO 5% gel — Once-daily applications, to the randomized side of the face either left or right, of clindamycin and benzoyl peroxide (BPO) 5% gel.
  Other Names: Duac Topical Gel
  Arms: Clindamycin and BPO 5% gel
Drug: Clindamycin phosphate and benzoyl peroxide 2.5% gel. — Once daily application of clindamycin phosphate and benzoyl peroxide (BPO) 2.5% gel
  Other Names: ACANYA Gel
  Arms: Clindamycin phosphate and BPO 2.5% gel

SUMMARY:
This is a single-blind (blinded expert grader) study that will enroll 25-30 healthy volunteers without facial acne. On 1 side of the face, the subject will apply 1 of the 2 test products, clindamycin and benzoyl peroxide 5% or clindamycin phosphate and benzoyl peroxide 2.5% and the other side of the face will remain non-treated to serve as a control.

DETAILED DESCRIPTION:
This is a single-blind (blinded expert grader), parallel group, randomized, half-face study being conducted at one clinical site. On 1 side of the face, the subject will apply 1 of the 2 test products, clindamycin and benzoyl peroxide 5%) or clindamycin and benzoyl peroxide 2.5%) and the other side of the face will remain non-treated to serve as a control. Approximately 25-30 male and female healthy subjects without facial acne, aged 18 to 45, will be randomly assigned to each product.

The eligible subjects (screened 3 days prior to randomization) who qualify will be entered into a 2-week treatment phase. The once-daily applications for the clindamycin and benzoyl peroxide 5%and clindamycin phosphate and benzoyl peroxide 2.5%) will be supervised at the site, Monday through Friday of each week. Subjects will apply the study product at home on Saturdays and Sundays and record the times of application on a diary card.

A blinded expert grader will rate comparative product tolerance in terms of erythema and dryness on each week day (excluding Saturdays and Sundays) during the study before study product is applied.

Instruments will be used to measure transepidermal water loss (TEWL) to assess skin moisture in order to evaluate product mildness. Instrumentation measurements of skin surface conductance will be utilized to evaluate product performance in terms of level of skin hydration.

Subjects will complete questionnaires and all adverse events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed.
* Male and female subjects aged from 18 to 45 years at time of consent.
* Is willing to discontinue use of all facial products (other than the cleanser provided and makeup or razor and facial shave product) on the face for the 3 days before their baseline/day 0 visit and use only the provided facial products and their normal makeup or razor and facial shaving product for the duration of the study.
* Is willing to not change brands of makeup or razor and facial shave product during the study.
* Is willing to refrain from using any facial product on the face other than study products and their normal makeup or razor and facial shave product for the duration of the study.
* Able to complete the study and to comply with study instructions.
* Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product

Exclusion Criteria:

* Female subjects who are pregnant, trying to become pregnant, or breast feeding.
* Male subjects that have facial beards (mustache and/or goatee is acceptable).
* Is a Type I diabetic.
* Has active or chronic skin allergies.
* Has a history of acute or chronic disease that might interfere with, or increase the risk of study participation.
* Has participated in other facial studies in the preceding 30 days or other clinical studies in preceding 14 days.
* Had skin cancer treatment in preceding 12 months.
* Has damaged skin on facial areas (eg, from sunburn, tattoos, scars).
* Had any medical procedure (eg, laser resurfacing, chemical peels, plastic surgery) to facial areas in preceding 12 months.
* Had any cosmetic procedure (eg, microdermabrasion, etc.) to facial areas within 8 weeks of the baseline visit.
* Use of topical retinoids or related agents for the treatment of acne or photoaging in the preceding 6 months.
* Any dermatological disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's facial appearance.
* Has known sensitivities or allergies to cosmetics, soaps, fragrances, or any of the ingredients in the test products.
* Is currently going through menopause and experiencing hot flashes.
* Received any investigational drug within 30 days of study day 0 or who are scheduled to receive an investigational drug other than the study product during the study.
* Currently using any medication, which in the opinion of the investigator may affect the evaluation of the study product or place the subject at undue risk (including but not limited to asthma medications, oral steroids, rifampin, anticonvulsants, St. John's wart).
* Currently taking any topical or oral erythromycin-containing products.
* History of regional enteritis, ulcerative colitis, or antibiotic-associated colitis.
* Currently suffering from any disease or condition, which in the opinion of the investigator may affect the evaluation of the study product or place the subject at undue risk.
* Live in the same household as currently enrolled subjects.
* Employees of investigator/ clinical research organization (CRO) or Stiefel, a GSK Company involved in the study, or an immediate family member (partner, offspring, parents, siblings or sibling's offspring) of an employee involved in the study.
* Any other condition or factor the investigator or his duly assigned representative believes may affect the skin response or the interpretation of the test results.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- cyberDERM, Broomall, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 114546 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114546 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114546 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114546 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114546 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Clinical research center. Enrollment started: 11 Aug 2009 Last patient last visit: 1 Sep 2009
Pre-assignment Details: Subjects who met inclusion and exclusion criteria and are willing to participate in the study were required to undergo a 3-day screening period where they will stop the use of all facial products on their face. Subjects were required to use soap free cleanser for washing their face and may apply their normal makeup.
Groups:
- Clindamycin and BPO 5% Gel: Once-daily applications, to the randomized side of the face either left or right, of clindamycin and benzoyl peroxide 5% gel.
- Clindamycin Phosphate and BPO 2.5% Gel: Once Daily application of clindamycin phosphate and benzoyl peroxide 2.5% gel.
Period: Overall Study
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Started | 17 | 19
Completed | 16 | 19
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 16 | 19 | 35
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 15 | 26
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Erythema (Redness)
Description: Compare tolerability of clindamycin and benzoyl peroxide (BPO) 5% and clindamycin phosphate and benzoyl peroxide 2.5% using visual assessments by an independent blinded grader.
  Erythema (redness) was evaluated using the following scale:
  Erythema Grade Description 0 = None 2 = Mild erythema 4 = Moderate confluent erythema 6 = Marked erythema with some edema 8 = Marked erythema, edema, possible erosion
Time Frame: 14 days
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
units on a scale
  Day 0 | 0.94 (0.83) | 1.05 (0.78)
  Day 1 | 1.42 (1.32) | 1.24 (.70)
  Day 2 | 1.45 (1.18) | 1.49 (1.33)
  Day 3 | 1.27 (.96) | 1.36 (1.14)
  Day 6 | 1.55 (1.15) | 1.87 (1.23)
  Day 7 | 1.72 (1.14) | 1.88 (1.25)
  Day 8 | 1.39 (.86) | 1.70 (1.38)
  Day 9 | 1.38 (1.00) | 1.82 (1.38)
  Day 10 | 1.78 (1.26) | 1.72 (1.18)
  Day 13 | 1.34 (1.03) | 1.82 (1.44)
  Day 14 | 1.51 (1.06) | 1.82 (1.18)
Statistical Analysis 1: Comparison: Clindamycin and BPO 5% Gel vs Clindamycin Phosphate and BPO 2.5% Gel; Test type: Superiority or Other; p > 0.05, Kruskal-Wallis

2. Secondary Outcome: Skin Moisture and Hydration
Description: To assess skin moisture and hydration using transepidermal water loss (TEWL). Results are measured on a continuous scale as grams per meters squared (m^2) per hour. Higher values indicate greater water loss/ lower skin moisture levels.
  Evaporative water loss measurements provide an instrumental assessment of skin barrier function(one of the layers of the skin. Damage leads to a disruption of the barrier that is accompanied by elevated water loss rates and affects skin moisture and hydration.
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: grams/m^2/hour
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
grams/m^2/hour
  Day 0 | 10.82 (4.15) | 9.71 (3.14)
  Day 3 | 11.98 (4.18) | 10.84 (3.46)
  Day 7 | 13.01 (3.16) | 11.36 (2.91)
  Day 14 | 13.94 (4.10) | 13.59 (4.68)
Statistical Analysis 1: Comparison: Clindamycin and BPO 5% Gel vs Clindamycin Phosphate and BPO 2.5% Gel; Test type: Superiority or Other; p > 0.05, Dunn's Multiple Comparisons Test

3. Primary Outcome: Skin Dryness
Description: Visual Dryness was evaluated using the following scale:
  Grade 0 = None 2 = Slight flaking 4 = Moderate flaking/scaling 6 = Marked scaling / slight fissuring 8 Severe scaling, fissuring
Time Frame: 14 days
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
units on a scale
  Day 0 | 0.06 (0.24) | 0.05 (0.23)
  Day 1 | 0.05 (0.05) | 0.15 (0.30)
  Day 2 | 0.05 (0.05) | 0.37 (0.66)
  Day 3 | 0.27 (0.55) | 0.22 (0.37)
  Day 6 | 0.29 (0.55) | 0.24 (0.53)
  Day 7 | 0.32 (0.54) | 0.15 (0.45)
  Day 8 | 0.40 (0.59) | 0.15 (0.32)
  Day 9 | 0.35 (0.56) | 0.15 (0.30)
  Day 10 | 0.47 (1.04) | 0.36 (0.99)
  Day 13 | 0.76 (1.33) | 0.28 (0.46)
  Day 14 | 0.62 (1.05) | 0.31 (0.54)
Statistical Analysis 1: Comparison: Clindamycin and BPO 5% Gel vs Clindamycin Phosphate and BPO 2.5% Gel; Test type: Superiority or Other; p > 0.05, Kruskal-Wallis

4. Secondary Outcome: Changes in the Skin Surface Hydration
Description: The ability of an alternating current to flow through the stratum corneum is an indirect measure of its water content. The value recorded is expressed in microsiemens. Higher values indicate greater levels of skin hydration.
  Test results were compared to measurements from the other side of the face, which was not treated instead of referring to a normal range. A normal range does not exist for this measurement. Instead, the non-treated side of the face was used as a control to determine the normal level of skin hydration.
Time Frame: 14 days
Population: ITT
Measure: Mean (Standard Deviation); unit: microsiemens
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
microsiemens
  Day 0 | 546.40 (185.75) | 478.02 (170.88)
  4 Hours Post 1st Treatment | 554.00 (202.94) | 430.78 (158.98)
  Day 3 | 572.39 (200.31) | 529.96 (124.88)
  Day 7 | 484.94 (212.56) | 413.51 (131.31)
  Day 14 | 361.59 (177.01) | 354.46 (144.06)
Statistical Analysis 1: Comparison: Clindamycin and BPO 5% Gel vs Clindamycin Phosphate and BPO 2.5% Gel; Test type: Superiority or Other; p > 0.05, Tukey-Kramer Multiple Comparisons Test

5. Secondary Outcome: Subject Tolerability - Burning
Description: At each visit, panelists were supplied a self-assessment questionnaire. Subjects were asked to evaluate burning, stinging, pain, and dryness in this questionnaire. Each symptom was rated with the following scale: 0 - None, 1 - Slight, 2 - Moderate, or 3 - Severe.
  The subjects completed this questionnaire prior to their daily application. The subjects used the time period (last 24 hours), from their last study application to the time they are administered this questionnaire for rating each symptom. The results for assessment of burning are presented here.
Time Frame: 2 weeks
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
units on a scale
  Day 0 | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.00 (0.00) | 0.00 (0.00)
  Day 2 | 0.00 (0.00) | 0.00 (0.00)
  Day 3 | 0.00 (0.00) | 0.00 (0.00)
  Day 6 | 0.00 (0.00) | 0.00 (0.00)
  Day 7 | 0.00 (0.00) | 0.00 (0.00)
  Day 8 | 0.00 (0.00) | 0.00 (0.00)
  Day 9 | 0.00 (0.00) | 0.00 (0.00)
  Day 10 | 0.00 (0.00) | 0.00 (0.00)
  Day 13 | 0.00 (0.00) | 0.00 (0.00)
  Day 14 | 0.00 (0.00) | 0.00 (0.00)

6. Secondary Outcome: Subject Tolerability - Stinging
Description: At each visit, panelists were supplied a self-assessment questionnaire. Subjects were asked to evaluate burning, stinging, and dryness in this questionnaire. Each symptom will be rated with the following scale: 0 - None,1 - Slight,2 - Moderate, or 3 - Severe.
  The subjects completed this questionnaire prior to their daily application. The subjects used the time period (last 24 hours), from their last study application to the time they are administered this questionnaire for rating each symptom. The results for assessment of stinging are presented here.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
units on a scale
  Day 0 | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.00 (0.00) | 0.00 (0.00)
  Day 2 | 0.06 (0.24) | 0.00 (0.00)
  Day 3 | 0.00 (0.00) | 0.05 (0.23)
  Day 6 | 0.00 (0.00) | 0.05 (0.23)
  Day 7 | 0.00 (0.00) | 0.00 (0.00)
  Day 8 | 0.00 (0.00) | 0.00 (0.00)
  Day 9 | 0.00 (0.00) | 0.00 (0.00)
  Day 10 | 0.00 (0.00) | 0.05 (0.23)
  Day 13 | 0.00 (0.00) | 0.00 (0.00)
  Day 14 | 0.00 (0.00) | 0.11 (0.46)

7. Secondary Outcome: Subject Assessment - Dryness
Description: At each visit, panelists were supplied a self-assessment questionnaire. Subjects were asked to evaluate burning, stinging, and dryness in this questionnaire. Each symptom will be rated with the following scale: 0 - None, 1 - Slight, 2 - Moderate, or 3 - Severe.
  The subjects completed this questionnaire prior to their daily application. The subjects used the time period (last 24 hours), from their last study application to the time they are administered this questionnaire for rating each symptom. The results for assessment of dryness are presented here.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
units on a scale
  Day 0 | 0.00 (0.00) | 0.26 (0.56)
  Day 1 | 0.00 (0.00) | 0.26 (0.56)
  Day 2 | 0.00 (0.00) | 0.21 (0.54)
  Day 3 | 0.00 (0.00) | 0.11 (0.46)
  Day 6 | 0.06 (0.24) | 0.11 (0.32)
  Day 7 | 0.12 (0.49) | 0.21 (0.54)
  Day 8 | 0.12 (0.49) | 0.16 (0.50)
  Day 9 | 0.2 (0.5) | 0.16 (0.50)
  Day 10 | 0.24 (0.56) | 0.16 (0.50)
  Day 13 | 0.35 (0.70) | 0.16 (0.50)
  Day 14 | 0.24 (0.56) | 0.21 (0.63)

8. Secondary Outcome: Subject Assessment - Roughness
Description: At each visit, panelists were supplied a self-assessment questionnaire. Subjects were asked to evaluate burning, stinging, roughness, and dryness in this questionnaire. Each symptom will be rated with the following scale: 0 - None, 1 - Slight, 2 - Moderate, or 3 - Severe.
  The subjects completed this questionnaire prior to their daily application. The subjects used the time period (last 24 hours), from their last study application to the time they are administered this questionnaire for rating each symptom. The results for assessment of roughness are presented here.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
units on a scale
  Day 0 | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.00 (0.00) | 0.05 (0.23)
  Day 2 | 0.00 (0.00) | 0.00 (0.00)
  Day 3 | 0.00 (0.00) | 0.00 (0.00)
  Day 6 | 0.06 (0.24) | 0.00 (0.00)
  Day 7 | 0.06 (0.24) | 0.00 (0.00)
  Day 8 | 0.06 (0.24) | 0.05 (0.23)
  Day 9 | 0.18 (0.53) | 0.05 (0.23)
  Day 10 | 0.12 (0.49) | 0.05 (0.23)
  Day 13 | 0.00 (0.00) | 0.05 (0.23)
  Day 14 | 0.00 (0.00) | 0.05 (0.23)

9. Secondary Outcome: Subject Assessment - Pain
Description: At each visit, panelists were supplied a self-assessment questionnaire, which included assessment of pain.
  Subjects were asked to evaluate burning, stinging, pain, and dryness in this questionnaire. Each symptom will be rated with the following scale: 0 - None, 1 - Slight, 2 - Moderate, or 3 - Severe.
  The subjects completed this questionnaire prior to their daily application. The subjects used the time period (last 24 hours), from their last study application to the time they are administered this questionnaire for rating each symptom. The results for assessment of pain are presented here.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
units on a scale
  Day 0 | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.00 (0.00) | 0.00 (0.00)
  Day 2 | 0.00 (0.00) | 0.00 (0.00)
  Day 3 | 0.00 (0.00) | 0.00 (0.00)
  Day 6 | 0.00 (0.00) | 0.00 (0.00)
  Day 7 | 0.00 (0.00) | 0.00 (0.00)
  Day 8 | 0.00 (0.00) | 0.00 (0.00)
  Day 9 | 0.00 (0.00) | 0.00 (0.00)
  Day 10 | 0.00 (0.00) | 0.00 (0.00)
  Day 13 | 0.00 (0.00) | 0.00 (0.00)
  Day 14 | 0.00 (0.00) | 0.00 (0.00)

10. Secondary Outcome: Subject Assessment - Crusting
Description: At each visit, panelists were supplied a self-assessment questionnaire. Subjects were asked to evaluate crusting, burning, stinging, and dryness in this questionnaire. Each symptom will be rated with the following scale: 0 - None, 1 - Slight, 2 - Moderate, or 3 - Severe.
  The subjects completed this questionnaire prior to their daily application. The subjects used the time period (last 24 hours), from their last study application to the time they are administered this questionnaire for rating each symptom. The results for assessment of crusting are presented here.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
units on a scale
  Day 0 | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.00 (0.00) | 0.00 (0.00)
  Day 2 | 0.00 (0.00) | 0.00 (0.00)
  Day 3 | 0.00 (0.00) | 0.00 (0.00)
  Day 6 | 0.00 (0.00) | 0.00 (0.00)
  Day 7 | 0.00 (0.00) | 0.00 (0.00)
  Day 8 | 0.00 (0.00) | 0.00 (0.00)
  Day 9 | 0.00 (0.00) | 0.00 (0.00)
  Day 10 | 0.00 (0.00) | 0.00 (0.00)
  Day 13 | 0.00 (0.00) | 0.00 (0.00)
  Day 14 | 0.00 (0.00) | 0.00 (0.00)

11. Secondary Outcome: Subject Assessment - Blistering
Description: At each visit, panelists were supplied a self-assessment questionnaire. Subjects were asked to evaluate blistering, burning, stinging, and dryness in this questionnaire. Each symptom will be rated with the following scale: 0 - None, 1 - Slight, 2 - Moderate, or 3 - Severe.
  The subjects completed this questionnaire prior to their daily application. The subjects used the time period (last 24 hours), from their last study application to the time they are administered this questionnaire for rating each symptom. The results for assessment of blistering are presented here.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
units on a scale
  Day 0 | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.00 (0.00) | 0.00 (0.00)
  Day 2 | 0.00 (0.00) | 0.00 (0.00)
  Day 3 | 0.00 (0.00) | 0.00 (0.00)
  Day 6 | 0.00 (0.00) | 0.00 (0.00)
  Day 7 | 0.00 (0.00) | 0.00 (0.00)
  Day 8 | 0.00 (0.00) | 0.00 (0.00)
  Day 9 | 0.00 (0.00) | 0.00 (0.00)
  Day 10 | 0.00 (0.00) | 0.00 (0.00)
  Day 13 | 0.00 (0.00) | 0.00 (0.00)
  Day 14 | 0.00 (0.00) | 0.00 (0.00)

12. Secondary Outcome: Subject Assessment - Oiliness
Description: At each visit, panelists were supplied a self-assessment questionnaire. Subjects were asked to evaluate oiliness, burning, stinging, and dryness in this questionnaire. Each symptom will be rated with the following scale: 0 - None, 1 - Slight, 2 - Moderate, or 3 - Severe.
  The subjects completed this questionnaire prior to their daily application. The subjects used the time period (last 24 hours), from their last study application to the time they are administered this questionnaire for rating each symptom. The results for assessment of oiliness are presented here.
Time Frame: 2 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Number analyzed (Participants) | 17 | 19
units on a scale
  Day 0 | 0.18 (0.53) | 0.16 (0.37)
  Day 1 | 0.18 (0.39) | 0.05 (0.23)
  Day 2 | 0.06 (0.24) | 0.00 (0.00)
  Day 3 | 0.12 (0.33) | 0.11 (0.46)
  Day 6 | 0.06 (0.24) | 0.00 (0.00)
  Day 7 | 0.06 (0.24) | 0.00 (0.00)
  Day 8 | 0.06 (0.24) | 0.00 (0.00)
  Day 9 | 0.06 (0.24) | 0.00 (0.00)
  Day 10 | 0.00 (0.00) | 0.00 (0.00)
  Day 13 | 0.00 (0.00) | 0.00 (0.00)
  Day 14 | 0.00 (0.00) | 0.00 (0.00)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Any study product-related AEs ongoing at the end of the treatment period would be followed until resolved, the condition stabilized, the events are otherwise explained, or the subject was lost to follow-up. In addition, all SAEs would have been followed until resolution as previously stated for study product-related AEs.
Arm/Group | Clindamycin and BPO 5% Gel | Clindamycin Phosphate and BPO 2.5% Gel
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 2/17 | 3/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clindamycin and BPO 5% Gel (N=17) | Clindamycin Phosphate and BPO 2.5% Gel (N=19)
Headache (Nervous system disorders) | 2 (2) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No